CLINICAL TRIAL: NCT03690596
Title: Personalized Smoking Relapse Prevention Delivered in Real-Time Via Just-in-Time-Adaptive Interventions
Brief Title: Smoking Relapse Prevention Via Just-in-Time-Adaptive Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meharry Medical College (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00061239; K23DA041616 (NIH)
Record Dates: First submitted 2018-09-24; First posted 2018-10-01 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy; Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NRT + QuitBuddy (Experimental): This smartphone app will identify high-risk situations through real-time EMA data collected before and during a quit attempt. One week of pre-quit smoking behaviors will be integrated with passively sensed GPS data to create hotspot maps. Hotspot maps will provide interactive visualizations of relapse risk. GPS triggered NRT/behavioral prompts will occur when participants come within 50m from the centroid of a hotspot.
  Interventions: Other: NRT + QuitBuddy
- NRT + QuitBuddy-Recall (Experimental): This smartphone app will identify high-risk situations through retrospective recall of locations where the patient typically smoked. Hotspot maps will provide interactive visualizations of relapse risk. GPS triggered NRT/behavioral prompts will occur when participants come within 50m from the centroid of a hotspot.
  Interventions: Other: NRT + QuitBuddy-Recall
- NRT Control (treatment as usual) (Active Comparator): Standard Care Control is intended to approximate the real-world experience where smokers obtain over-the-counter NRT and, after brief instructions at the outset (~1 lozenge per hour, during cravings, and <20 per day), determine usage for themselves.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: NRT + QuitBuddy — QuitBuddy treatment app and 1 month supply of 4 mg nicotine lozenge
  Arms: NRT + QuitBuddy
Other: NRT + QuitBuddy-Recall — QuitBuddy-Recall treatment app and 1 month supply of 4 mg nicotine lozenge
  Arms: NRT + QuitBuddy-Recall
Other: Treatment as Usual — 1 month supply of 4 mg nicotine lozenge
  Arms: NRT Control (treatment as usual)

SUMMARY:
A small-scale randomized controlled trial (RCT) will pilot test a personalized JITAI designed to guide delivery of fast acting nicotine replacement therapy (NRT; lozenge) in real-time, to prevent smoking relapse. Specifically, a smartphone application (app), will integrate pre-quit smoking data with objective location data captured via global positioning system (GPS) to establish relapse risk (hotspot) algorithms. During a quit attempt, the GPS-enabled app (QuitBuddy) will detect proximity to hotspots and deliver NRT prompts, all of which will occur automatically and prior to exposure. Thus, QuitBuddy will optimize NRT use to prevent cue-provoked cravings known to undermine sustained abstinence, thereby repurposing this evidence-based cessation medication to promote relapse prevention. QuitBuddy will be tested against standard care (NRT with brief instructions). Two versions of QuitBuddy will be tested, which will differ only in how hotspot algorithms are derived: retrospectively from locations recalled at the onset of a quit attempt (QuitBuddy-Recall) or based on real-time EMA completed pre-quit (QuitBuddy).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* daily cigarette smoker of > 9 cigarettes/day for past year
* CO breath monitor detects > 10ppm
* literate in English
* willing to make a quit attempt in the next week with nicotine replacement therapy
* no plans to travel outside of a 100-mile radius of Charleston during the study

Exclusion Criteria:

* FDA contraindications for use of NRT:

  1. Pregnant
  2. Breastfeeding or planning to become pregnant
  3. Recent (past 3 months) cardiovascular trauma: MI, stroke
* current use (past 30 days) of alternative tobacco products or smoking cessation medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-04-16 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Abstinence from cigarettes | 12 Weeks
  Biochemically-verified smoking status (CO<6) obtained at 3-month follow-up

SECONDARY OUTCOMES:
Abstinence from cigarettes | 4 weeks
  Biochemically-verified smoking status (CO<6) obtained at 1-month follow-up
Abstinence from cigarettes | 1 week
  Biochemically-verified smoking status (CO<6) obtained at 1-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bryan W Heckman, PhD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States